CLINICAL TRIAL: NCT01467778
Title: A Phase I Study to Assess the Safety of Three Formulations of the Dermal Implant ELAPR in Healthy Subjects
Brief Title: Safety Study of Three Formulations of the Dermal Implant ELAPR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elastagen Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: ELAPR-P1
Record Dates: First submitted 2011-03-22; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Skin Conditions
Keywords: skin
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ELAPR001 (Active Comparator): Tropoelastin 0.1ml SC implant
  Interventions: Device: ELAPR
- ELAPR002 (Active Comparator): Tropoelastin 0.1ml SC implant
  Interventions: Device: ELAPR
- ELAPR003 (Active Comparator): Tropoelastin 0.1ml SC implant
  Interventions: Device: ELAPR
- Saline (Placebo Comparator): Normal Saline 0.9%
  Interventions: Device: ELAPR

INTERVENTIONS:
Device: ELAPR — ELAPR implant product is under development for mid to deep dermal implantation for the treatment of the symptoms of skin aging including the correction of moderate to sever facial wrinkles and folds, such as nasolabial folds and skin abnormalities such as scars.
  Other Names: Other Names:; Tropoelastin 0.1ml SC implant
Device: ELAPR — Implant area of the medial aspect of the upper arm along the posterior line of the bicep is to be selected where there are no pigmentations or moles. Injections will be marked with a tattoo and placed at 2 cm intervals. The order is to be from proximal to distal control, ELAPR001, ELAPR002, ELAPR003
  Other Names: Tropoelastin 0.1ml SC implant

SUMMARY:
This is a Phase I study to assess the safety of three formulations of the dermal implant ELAPR.

DETAILED DESCRIPTION:
A Phase I study to assess the safety of three formulations of the dermal implant ELAPR in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Good general health status

Exclusion Criteria:

* Clinically significant abnormalities of haematology or biochemistry testing
* Bleeding diathesis, anticoagulant drugs,thrombocytopenia or clinically significant prolonged APTT or PT
* Chronic use of aspirin, other non-steroidal antiinflammatory drugs or other anti-platelet agents
* History of keloid formation
* Systemic corticosteroids within last 12 weeks
* Diabetes or metabolic disorders
* Any serious medical condition which in the opinion of the investigator would have a strong possibility of requiring systemic corticosteroid medication
* Pregnancy/lactation
* A history of anaphylaxis or allergic reactions including any known hypersensitivity to Hyaluronic acid or lidocaine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability measured by the amount of adverse events and serious adverse events | 6 weeks
  To assess the safety and tolerability of a single course of intradermal injections of ELAPR when administered to healthy subjects by reported adverse events and serious adverse events

SECONDARY OUTCOMES:
Persistence | 6 weeks
  To determine implant persistence by histopathology and clinical observation

CONTACTS AND LOCATIONS:
Overall Officials: Carlos China, MBBS, Principal Investigator — Woolcock Institute of Medical Research
Locations (1):
- Woolcock Institute of Medical Research, Glebe, New South Wales, Australia